CLINICAL TRIAL: NCT05885529
Title: Added Value, Performance and Acceptance of the "GFAP-UCH-L1" Pair in the Evaluation of Subjects with Mild Traumatic Brain Injury (MTBI) At Intermediate Risk of Complications
Brief Title: Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin Carboxy-terminal Hydrolase L1 (UCH-L1) to Exclude Lesions Linked to Significant Traumatic Brain Injuries
Acronym: GUEST
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Collaborators: BioMérieux (Industry); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Clermont-Ferrand (Other); Hospices Civils de Lyon (Other); Poitiers University Hospital (Other); University Hospital, Angers (Other Government); Centre Hospitalier Universitaire de Nīmes (Other); Centre Hospitalier Universitaire de Nice (Other); Nantes University Hospital (Other); University Hospital, Montpellier (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Grenoble (Other); Fondation Hôpital Saint-Joseph (Other); CHU de Tours (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22-22
Record Dates: First submitted 2023-05-04; First posted 2023-06-02 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
Keywords: UCHL1; GFAP; CT scan
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample obtained at initial presentation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- consecutive participants in the 15 centers: adult patients with mild traumatic brain injury admitted within 12 hours after the trauma. No interventions, observational study
  Interventions: Other: UCH-L1 GFAP

INTERVENTIONS:
Other: UCH-L1 GFAP — measurment of UCH-L1 GFAP within 12 hours in adult patients after a mild traumatic brain injury

SUMMARY:
The goal of this observational study is to evaluate the performance of UCH-L1 and GFAP combined in patients with a mild traumatic brain injury. The main question :

• Does the combination of UCH-L1 and GFAP can exclude brain injuries detected with CT scan in the first twelve hours after a mild traumatic brain injury?

Participants will do the exams planed in routine care and :

* during the expected blood sampling an additional blood sample will be done,
* seven days after the discharge a call will be done by the investigator.

DETAILED DESCRIPTION:
Main study

The main study includes subjects presenting to the emergency department within 12 hours of mild traumatic brain injury with an intermediate risk of clinical worsening or intracranial lesions.

The participants have at least one of the following characteristics, as defined in the French recommendations

* > 65 years treated with anti-platelet agents
* Glasgow Score < 15 at two hours after the trauma if associated intoxication (alcohol, narcotic, psychotropic)
* Trauma with high kinetics (for information only: a risk mechanism (pedestrian knocked down by a motorized vehicle, ejection from a vehicle, fall from more than 3 steps (more than one meter), etc.),
* Amnesia of facts > 30 min before the trauma

The study includes clinical sites in France and Monaco. Participants have a blood sample and a brain scan as part of the care. The participation of subjects in the study will not influence their treatment.

Ancillary study The ancillary study uses qualitative research methodology to assess acceptance by physicians and patients of a biological test rather than a CT scan to exclude intracranial complication after mild traumatic brain injury.

The study will takes place in the emergency department of the Nice University Hospital Center (CHU of Nice). It will include 30 subjects: 15 subjects presenting to the emergency room for mild traumatic brain injury and included in the main protocol and 15 prescribing emergency physicians.

The participation of subjects in the study will not influence their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury defined by

  * Impact on the skull or the face AND OR
  * Acceleration / deceleration
* Glasgow Coma Scal 13, 14 or 15
* One of the following 4 criteria:

  * > 65 years treated with anti-platelet agent,
  * GCS < 15 two hours after the trauma if associated intoxication (alcohol, narcotic, psychotropic),
  * Trauma with high kinetics (for information only: a risk mechanism (pedestrian knocked down by a motorized vehicle, ejection from a vehicle, fall from more than 3 steps (more than one meter), etc.),
  * Amnesia of facts > 30 min before the trauma.
* Having a blood sample taken as part of care with a delay between the clinical event and the biological sample < 12 hours
* Having a CT-scan prescription as part of the MTBI evaluation
* Patient who signed an informed consent form

Exclusion Criteria:

* Person not affiliated or not benefiting from a health insurance scheme.
* Person under judicial protection.
* Person with restrictions of freedom or subject to Articles L.3212-1 and L.3213-1, and not included in Article L.1122-8 of the French CSP
* Blood collection time > 12 hours
* Subjects for which a scan would be carried out systematically, including:

  * GCS <13 (moderate or severe trauma),
  * congenital hemostasis disorders or patient on anti-coagulant treatment,
  * clinical signs evoking a fracture of the vault or the base of the skull,
  * more than one episode of vomiting,
  * post-traumatic convulsion,
  * focal neurological deficit.
* Obstacle to follow-up at D7
* Malignant melanomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects consulting in the emergency department within 12 hours following a mild traumatic brain injury at risk of complications meeting the inclusion and exclusion criteria listed in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
performance of UCH-L1 and GFAP combined to rule out intracranial complication after MTBI | during the first 12 hours
  Percentage of intracranial lesion excluded by UCH-L1 and GFAP combined, versus the CT scan, within the first 12 hours following a MTBI

SECONDARY OUTCOMES:
Performance of UCH-L1 and GFAP combined to rule out intracranial bleeding after MTBI | during the first 12 hours
  Percentage of intracranial bleeding excluded by UCH-L1 and GFAP alone or combined, versus the CT scan, within the first 12 hours following a MTBI
Performance of UCH-L1 and GFAP combined to rule out intracranial bleeding after MTBI | during the first 12 hours with a focus every 3 hours
  Percentage of intracranial lesion excluded by UCH-L1 and GFAP alone or combined, versus the CT scan, within the first 12 hours following a MTBI .
Comparation of UCH-L1 and GFAP combined or alone, to S100b protein (PS100b) | during the first 12 hours with a focus every 3 hours
  Percentage of intracranial complication identified by UCH-L1 and GFAP, alone or in combination, versus PS100b within the first 12 hours following a MTBI .
Predicted impact of using UCH-L1 and GFAP combined | day 7
  Variation of resource consumption by the use of UCH-L1 and GFAP
Performance of UCHL-1 and GFAP alone or combined to predict complications | during the first 7 days
  Percentage of complications avoided by the use of UCH-L1 and GFAP, alone or combined.

OTHER OUTCOMES:
ancillary outcome | Day 1
  Acceptability by a semi-directed interview of a new strategy integrating the use of biomarkers for the management of MTBI by patients and investigators

CONTACTS AND LOCATIONS:
Overall Officials: Pierre HAUSFATER, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (15):
- France (14):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Gabriel-Montpied - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital François Mitterrand - CHU de Dijon, Dijon
  - Hôpital Nord - CHU de Grenoble-Alpes, Grenoble
  - Hospices Civils de Lyon, Lyon
  - Hôpital Lapeyronie - CHU de Montpellier, Montpellier
  - Hôtel Dieu - CHU de Nantes, Nantes
  - Hôpital Pasteur CHU de Nice, Nice
  - Hôpital Carémeau - CHU de Nîmes, Nîmes
  - AP-HP Nord Lariboisière, Paris
  - AP-HP Sorbonne Université, site Pitié-Salpêtrière, Paris
  - Hôpital Saint-Joseph, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hôpital Trousseau - CHRU Tours, Tours
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No